CLINICAL TRIAL: NCT03954509
Title: Needs Assessment of Cancer Patients With Complementary and Alternative Medicines
Acronym: MAC'EVAL
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Hopital Antoine Beclere (Other)
Responsible Party: Sponsor
Other Study IDs: MAC'EVAL
Record Dates: First submitted 2018-08-10; First posted 2019-05-17 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Cancer; Chemotherapy Effect
Keywords: Complementary and Alternative Medicines
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- semi-structured interview: Screening and inclusion of patients hospitalized or seen in day hospital to conduct semi-structured interviews according to the interview grid. This interview schedule was established after review of the literature and identification of primary and secondary objectives.
  * Identification of key ideas through content analysis of the interviews conducted and based of the anchored theory.
  * This step is performed until the results are saturated (approximately 15 patients). The principle of saturation is based on the fact that from a threshold, the diversity of the elements collected decreases. Much more than an end signal, this principle is "a methodological guarantee" since it allows the possibility of comparing divergent or contradictory data and thus validating the data.
- questionnaires: * From the previous results: elaboration of a written questionnaire built according to the results obtained thanks to the previous interviews. In order to apply the simple correspondence factor analysis method, this questionnaire will be constructed on a Likert scale. The objective is twofold:
    1. to reduce the observer's bias by considering both the literature reviews but also the points of view of patients to develop the questionnaire;
    2. reach a larger patient population (more than 100 patients) compared to the previous qualitative analysis (15 patients planned), in order to generalize the results. This methodology combines both qualitative and quantitative study to minimize bias induced by both types of study.
  * Dissemination of the questionnaire and filling by the patient independently. The health professional who submitted the questionnaire will remain available to answer any questions the patient may have.

SUMMARY:
The chronic cancer status, multidisciplinary and ambulatory care, as well as the cumbersome effects of the disease and treatments, lead patients to consider other options than those offered by traditional medicine, such as alternative medicine and complementary (CAM)

DETAILED DESCRIPTION:
In order to put in place a policy on CAM based on the knowledge held by the patient and the health professionals, it is imperative to obtain and analyze the following information: why this type of medicine is used, what are its benefits, how does the patient get information and what are his sources, who practices them and how the patient perceives the place of the hospital and the various health professionals to develop and secure the use of CAM.

Our study will focus on CAM that can bring iatrogenic risk (phytotherapy, food supplements, acupuncture, traditional Chinese medicine, homeopathy, essential oils), and the following techniques: hypnosis and sophrology.

The study is carried out in two successive phases: the interview phase which will make it possible to obtain results to carry out the questionnaires phase. Patients who will be included in the interview phase will not participate in the questionnaire phase. Finally, patients who participate in the questionnaire phase will not have semi-structured interviews. They will only have to answer the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Woman and man over 18
* Francophone (speaking and reading French)
* Patient followed for the management of cancer, hospitalized or not, receiving or having already received a treatment cancer administered orally and / or systemically.

Exclusion Criteria:

* Patient who has not been treated for cancer with anticancer treatment
* Support in a palliative care service
* Refusal to participate in the study
* Patient under tutorship or curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is carried out in two successive phases: the interview phase which will make it possible to obtain results to carry out the questionnaires phase. Patients who will be included in the interview phase will not participate in the questionnaire phase. Finally, patients who participate in the questionnaire phase will not have semi-structured interviews. They will only have to answer the questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of the perception of patients regarding complementary and alternative medicines (CAM) in the management of cancer or its complications but also the place of different health professionals. | Time of inclusion
  This evaluation is carried out using a semi-directed interview, then a questionnaire

SECONDARY OUTCOMES:
Prevalence of CAM used in cancer patients | Time of inclusion
  Number of cancer patients that use CAM
Number of factors influencing the consumption of CAM | Time of inclusion
  e.g. age, sex, type of cancer, perpeptions of the CAM
Number of iatrogenic risks related to CAM and chemotherapy | Time of inclusion
  CAM used by cancer patients and their chemotherapy
Number of the CAM supply sources | Time of inclusion
  e.g community pharmacies, supermarket, internet)
Number of the information sources used by patients | Time of inclusion
  questionnaire (eg internet, health professionals, TV)
Identification of the roles of health professionals in the patient's treatment process to help secure information about CAM | Time of inclusion
  questionnaire (eg health professionals,roles)

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Bernstein BJ, Grasso T. Prevalence of complementary and alternative medicine use in cancer patients. Oncology (Williston Park). 2001 Oct;15(10):1267-72; discussion 1272-8, 1283. PMID 11702957
- [Result] Naja F, Anouti B, Shatila H, Akel R, Haibe Y, Tfayli A. Prevalence and Correlates of Complementary and Alternative Medicine Use among Patients with Lung Cancer: A Cross-Sectional Study in Beirut, Lebanon. Evid Based Complement Alternat Med. 2017;2017:8434697. doi: 10.1155/2017/8434697. Epub 2017 Aug 24. PMID 28912824
- [Result] Ernst E, Cassileth BR. The prevalence of complementary/alternative medicine in cancer: a systematic review. Cancer. 1998 Aug 15;83(4):777-82. doi: 10.1002/(sici)1097-0142(19980815)83:43.0.co;2-o. PMID 9708945
- [Result] Horneber M, Bueschel G, Dennert G, Less D, Ritter E, Zwahlen M. How many cancer patients use complementary and alternative medicine: a systematic review and metaanalysis. Integr Cancer Ther. 2012 Sep;11(3):187-203. doi: 10.1177/1534735411423920. Epub 2011 Oct 21. PMID 22019489
- [Result] Garland SN, Valentine D, Desai K, Li S, Langer C, Evans T, Mao JJ. Complementary and alternative medicine use and benefit finding among cancer patients. J Altern Complement Med. 2013 Nov;19(11):876-81. doi: 10.1089/acm.2012.0964. Epub 2013 Jun 18. PMID 23777242
- [Result] Samuels N, Ben-Arye E, Maimon Y, Berger R. Unmonitored use of herbal medicine by patients with breast cancer: reframing expectations. J Cancer Res Clin Oncol. 2017 Nov;143(11):2267-2273. doi: 10.1007/s00432-017-2471-x. Epub 2017 Jun 30. PMID 28667389
- [Result] Ben-Arye E, Samuels N, Goldstein LH, Mutafoglu K, Omran S, Schiff E, Charalambous H, Dweikat T, Ghrayeb I, Bar-Sela G, Turker I, Hassan A, Hassan E, Saad B, Nimri O, Kebudi R, Silbermann M. Potential risks associated with traditional herbal medicine use in cancer care: A study of Middle Eastern oncology health care professionals. Cancer. 2016 Feb 15;122(4):598-610. doi: 10.1002/cncr.29796. Epub 2015 Nov 24. PMID 26599199
- [Result] Richardson MA, Sanders T, Palmer JL, Greisinger A, Singletary SE. Complementary/alternative medicine use in a comprehensive cancer center and the implications for oncology. J Clin Oncol. 2000 Jul;18(13):2505-14. doi: 10.1200/JCO.2000.18.13.2505. PMID 10893280
- [Result] Sparber A, Bauer L, Curt G, Eisenberg D, Levin T, Parks S, Steinberg SM, Wootton J. Use of complementary medicine by adult patients participating in cancer clinical trials. Oncol Nurs Forum. 2000 May;27(4):623-30. PMID 10833691
- [Result] Cassileth BR, Schraub S, Robinson E, Vickers A. Alternative medicine use worldwide: the International Union Against Cancer survey. Cancer. 2001 Apr 1;91(7):1390-3. doi: 10.1002/1097-0142(20010401)91:73.0.co;2-c. PMID 11283941
- [Result] Patterson RE, Neuhouser ML, Hedderson MM, Schwartz SM, Standish LJ, Bowen DJ, Marshall LM. Types of alternative medicine used by patients with breast, colon, or prostate cancer: predictors, motives, and costs. J Altern Complement Med. 2002 Aug;8(4):477-85. doi: 10.1089/107555302760253676. PMID 12230908
- [Result] Swisher EM, Cohn DE, Goff BA, Parham J, Herzog TJ, Rader JS, Mutch DG. Use of complementary and alternative medicine among women with gynecologic cancers. Gynecol Oncol. 2002 Mar;84(3):363-7. doi: 10.1006/gyno.2001.6515. PMID 11855870
- [Result] Molassiotis A, Panteli V, Patiraki E, Ozden G, Platin N, Madsen E, Browall M, Fernandez-Ortega P, Pud D, Margulies A. Complementary and alternative medicine use in lung cancer patients in eight European countries. Complement Ther Clin Pract. 2006 Feb;12(1):34-9. doi: 10.1016/j.ctcp.2005.09.007. Epub 2005 Nov 14. PMID 16401528
- [Result] Frenkel M, Cohen L. Effective communication about the use of complementary and integrative medicine in cancer care. J Altern Complement Med. 2014 Jan;20(1):12-8. doi: 10.1089/acm.2012.0533. Epub 2013 Jul 17. PMID 23863085
- [Result] Blodt S, Mittring N, Schutzler L, Fischer F, Holmberg C, Horneber M, Stapf A, Witt CM. A consultation training program for physicians for communication about complementary medicine with breast cancer patients: a prospective, multi-center, cluster-randomized, mixed-method pilot study. BMC Cancer. 2016 Nov 4;16(1):843. doi: 10.1186/s12885-016-2884-y. PMID 27809814
- [Result] Fong YK, Marihart S, Harik M, Djavan B. Preventing progression in men with mild symptoms of benign prostatic hyperplasia: a potential role for phytotherapy. Rev Urol. 2004 Fall;6(4):187-92. PMID 16985600
- [Result] Kim SW. Phytotherapy: emerging therapeutic option in urologic disease. Transl Androl Urol. 2012 Sep;1(3):181-91. doi: 10.3978/j.issn.2223-4683.2012.05.10. PMID 26816707